CLINICAL TRIAL: NCT00698542
Title: A Validation of a Patient Safety Screening Tool for Sepsis
Brief Title: Evaluation of the Patient Safety Screening Tool (PSST) for Sepsis
Status: Terminated | Type: Observational
Why Stopped: The study design failed and the data was not able to be analyzed.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, John Allan Barwis, Asssistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 80093
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Sepsis
Keywords: PSST; sepsis; Neuro Care Unit; Surviving Sepsis Campaign; SSC
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients in the NCU at VUH

SUMMARY:
The Patient Safety Screening Tool (PSST) for Sepsis solution is a tool to assist with the early detection of Sepsis and management of the administration of bundle packages as defined by the Institute for Healthcare Improvement (IHI). This web based application relies on integration with bedside medical equipment (BME) data as well as Lab and Registration data so that clinical workflow items can be automated in the fight against Sepsis.

DETAILED DESCRIPTION:
The workflow that is automated by the PSST for Sepsis solution is tightly integrated with Registration, Bedside Monitoring Equipment (BME), and Lab data. As patients arrive in the unit, workflow activities are started with patient context. Typical implementations of the IHI guidelines for Sepsis screening dictate that patients are rescreened on regular intervals to detect Sepsis. The PSST for Sepsis solution will monitor Lab and BME data stores and continually update the screening forms for a particular patient. It will also alert clinicians when a manual screen is required in the Microsoft InfoPath form. The constant screening loop is managed by the PSST for Sepsis solution and will continue to run until the patient screens positive for Severe Sepsis, or moves to the next workflow of auditing a patient with Sever Sepsis.

When patients reach a state of "positive screen" (either manually, or through the automated data monitors) the PSST for Sepsis solution will move this patient from a screening workflow to an auditing workflow automatically. The PSST for Sepsis solution will then monitor the treatment process through Microsoft InfoPath form posts and alert clinicians when treatment goals have not been met. After a successful auditing process and completion of the 6 and 24 hour bundles, the patient will be placed back into a screening workflow. The end result is that patients will remain in a screening/auditing workflow loop until the patient is discharged from the unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are hospitalized in the Neuro Care Unit (NCU)
* Patients that are hospitalized in the Vanderbilt Burn Center
* Patients must be > 18 years of age

Exclusion Criteria:

* Patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be located in the 22 bed Vanderbilt University Medical Center Neuro Care Unit (NCU). Every patient will be screened for sepsis according to the following workflow upon admission to the NCU. The patient population of the NCU is generally bimodal; the first group consists of post-operative patients with an average length of stay of three to five days. The second group consists of subarachnoid hemorrhage patients with an average length of stay of 45 days.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Demonstrate a reduction in time to detection of sepsis using the PSST Alert System | 6 and 24 hours

SECONDARY OUTCOMES:
Determine the accuracy of the PSST Alert System | 6 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: John A Barwise, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt University Medical Center Department of Anesthesiology — http://www.vandydreamteam.com